CLINICAL TRIAL: NCT05934370
Title: The Duke-Reinvestment Partners Community Collaborative (DRC)- Healthy Homes
Acronym: DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113089
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Other): Participants will receive an intervention kit that will include two at-home visits and the following products: child bedroom HEPA-air purifier, HEPA upright vacuum, hypoallergenic dust-mite cover for child's mattress and pillow covers; Non-toxic household cleaning products and non-toxic pest/rodent traps.
  Interventions: Other: Home-Based Environmental Interventions (HEI)

INTERVENTIONS:
Other: Home-Based Environmental Interventions (HEI) — Housing Specialist will conduct an environmental home assessment to identify asthma triggers.
  • The participant will receive the following Breath Easy at Home Kit Products:
  * HEPA filtered upright vacuum cleaner
  * HEPA-filtered air purifier
  * Hypoallergenic latex free mattress and pillow covers
  * Healthier household cleaners
  * Non-toxic pest control devices for rodent control
  * Safe products to locate and kill roaches.

SUMMARY:
The goal of this open-label, single arm home intervention feasibility study is to improve quality of life for children ages 4-16 years with asthma.

The main questions it aims to answer are:

* How can Home-Based Environmental Interventions (HEI) improve home air-quality problems in the home?
* How can HEI improve asthma outcomes in children?

Participants will be receiving HEI and completing asthma surveys.

DETAILED DESCRIPTION:
All participants will receive an Intervention Kit, which could help with reducing environmental exposures. Participants will be monitored closely with up to 2 clinic visits, 2 home visits and up to 4 phone call visits. During the home visits, a study team will ask questions about your home and asthma, conduct home assessments, and provide training on use of the home kit.

Participants may benefit from participation in this study through Home-Based Environmental Interventions by improving home air-quality and asthma outcomes. Study duration is approximately 24-30 weeks with 8 weeks of intervention, which includes baseline interview, questionnaires, spirometry testing, and participants receiving an Intervention Kit.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian has provided informed consent (child has provided assent if needed)
* 4-16 years of age with medical provider -diagnosed asthma
* Evidence of recent poor asthma control, defined as either:

  1. Asthma exacerbation requiring systemic steroids within 3 month of consent OR
  2. ACQ6 > 1.0; or ACT/cACT ≤ 19 during ambulatory visit within 3 months of consent
* Family lives in one of the following Central NC counties: Alamance, Chatham, Durham, Franklin, Granville, Johnston, Lee, Orange, Person, Vance, or Wake counties
* Family is not planning to move out of one of the approved counties accessible to Reinvestment Partners in the next 6 months

Exclusion Criteria:

* Lack of informed consent
* Any major chronic illness that in the opinion of the Principal Investigator (PI) would interfere with participation in the intervention or completion of the study procedures
* Inability to complete baseline measurements in a satisfactory manner according to the judgment of the research coordinator or PI
* Parent/Caregiver unable to consent in English or Spanish
* Sensitivity or allergy to silicone

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Week 10
  A measure of satisfaction by distributing a satisfaction survey to each patient and caregiver
Caregiver Satisfacation Survey | Week 10
  A measure of satisfaction by distributing a satisfaction survey to each patient and caregiver
Change in Air -Quality Index | Week 4, Week 10
  Air-quality index assessments will include: PM2.5, PM10, total VOC's, formaldehyde, carbon dioxide, Air Quality Index) in child's room and main living room using the Temtop M10, Temptop 2000C, and HEPA purifier air quality monitor.
Asthma healthcare utilization measured by number of clinic visits needed | Through study completion, an average of 24 weeks
  Determine ongoing need for healthcare utilization for participant's asthma
Asthma healthcare utilization measured by number of Emergency Department visits | Through study completion, an average of 24 weeks
  Determine ongoing need for healthcare utilization for participant's asthma
Asthma healthcare utilization measured by number of urgent care visits | Through study completion, an average of 24 weeks
  Determine ongoing need for healthcare utilization for participant's asthma
Asthma healthcare utilization measured by number of hospitalizations | Through study completion, an average of 24 weeks
  Determine ongoing need for healthcare utilization for participant's asthma

SECONDARY OUTCOMES:
Study Completion | Through study completion, an average of 24 weeks
  Study completion will be measured when 30 participants enroll and complete the intervention
Change in Air Quality of Formaldehyde measured by a Temtop M10 | Week 8
  The Temtop M10 will measure the amount of Formaldehyde in the home
Change in Air Quality of Particulate Matter (PM) measured by a Temtop M10 | Week 8
  The Temtop M10 will measure the amount of Particulate Matter (PM) 2.5 in the home
Change in Air Quality of TVOC measured by a Temtop M10 | Week 8
  The Temtop M10 will measure the amount of TVOC in the home
Change in Air Quality measured by a Temtop M10 | Week 8
  The Temtop M10 will measure the air quality in the home
Air Quality changes of Particulate Matter (PM) 2.5 measured by a Temtop M2000c | Week 8
  The Temtop M2000c will measure the Particulate Matter (PM)2.5
Air Quality changes of particles measured by a Temtop M2000c | Week 8
  The Temtop M2000c will measure the number of particles in the home
Air Quality changes of carbon dioxide measured by a Temtop M2000c | Week 8
  The Temtop M2000c will measure the amount of carbon dioxide in the home
Air Quality changes of particulate matter (PM 10) measured by a Temtop M2000c | Week 8
  The Temtop M2000c will measure the amount of particulate matter (PM 10) in the home
Air Quality changes measured by patient's air purifier | Week 8
  The patient's air purifier will measure the air quality index in the home
Measurement of lung function | Week 10
  Lung function will be measure by spirometry
Asthma Symptoms measured by the Asthma Control Questionnaire (ACQ 6) | Week 10
  The Asthma Control Questionnaire (ACQ 6) is a 6 question self-report measure of asthma symptoms over the prior week. Items are rated on a sale ranging from 0 (never interferes with daily life) to 6 (interferes very severely with daily life). Higher scores indicate a worse outcome than lower scores.
Asthma symptoms measured by the Asthma Control Test (ACT or cACT) | Week 10
  The Asthma Control Test (ACT or cACT) is a 5 question self-report measure of asthma symptoms over the prior four weeks. Items are rated on a scale ranging from 1 (All of the time) to 5 (none of the time). Lower scores indicate a worse outcome than higher scores.
Asthma symptoms measured by the Duke Asthma Score (DAS) | Week 10
  The Duke Asthma Score (DAS) is a 6 question self-report measure of asthma symptoms over the prior month. Items are rated on a scale ranging from 0 (never) to 4 (every day). Higher scores indicate a worse outcome than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No